CLINICAL TRIAL: NCT06690840
Title: A Phase II Study of Atezolizumab, Vinorelbine and Weekly Cyclophosphamide as T-cell Activators in First Line Metastatic Triple Negative Breast Cancer Patients Pre-treated With Anti-PD-L1/PD-1
Brief Title: Atezolizumab and Chemotherapy Treatment as T-cell Activators in Metastatic Triple Negative Breast Cancer Patients
Acronym: AZALEA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UID 2686
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; PD-L1-positive; Locally advanced or metastatic breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — atezolizumab; Cyclophosphamide; Vinorelbine

STUDY DESIGN:
Intervention Model Description: Open-label, phase II, single arm, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab plus Cyclophosphamide and Vinorelbine (Experimental): Atezolizumab 840 mg intravenous (IV) on Days 1 and 15 of every 28-day cycle in combination with Cyclophosphamide 300 mg/m2 IV on Days 1 ,8,15, 21 of every 28-day cycle and Vinorelbine 30 mg per os (PO) on Days 1, 3, 5 every week of every 28-day cycle
  Interventions: Drug: Atezolizumab in combination with Cyclophosphamide and Vinorelbine

INTERVENTIONS:
Drug: Atezolizumab in combination with Cyclophosphamide and Vinorelbine — Patients will receive Atezolizumab in combination with Cyclophosphamide and Vinorelbine in 28-day cycles

SUMMARY:
Triple-negative breast cancer (TNBC) is among the most aggressive and lethal types of breast cancer, and currently available therapies have an unsatisfactory impact on patients' survival.

The primary aim of this clinical trial is to evaluate efficacy in terms of Overall Response Rate (ORR) of atezolizumab plus cyclophosphamide and vinorelbine in first line patients with unresectable locally advanced or metastatic TNBC patients, previously treated with anti-programmed cell death ligand-1 (PD-L1) or anti-programmed cell death-1 (PD-1) - containing regimens, in the neoadjuvant/adjuvant setting.

DETAILED DESCRIPTION:
TNBC is among the most aggressive and lethal types of breast cancer, and currently available therapies have an unsatisfactory impact on patients' survival.

The association of checkpoint inhibitors (CIs) such as anti-PD-L1 with chemotherapy has shown some encouraging results in randomized clinical trials enrolling TNBC patients either in the early (neo-adjuvant) or in the advanced/metastatic setting, but there has been no clear evidence of what should be considered the best chemotherapy backbone to be associated with CIs.

What could be considered the most promising combinatorial regimen of chemotherapy plus anti-PDL1 was defined using two complementary TNBC models at the preclinical level. The present phase II study will investigate overall response rate (ORR) as primary endpoint in first line metastatic TNBC patients treated with this investigational combination comprising atezolizumab (A) Vinorelbine (V), and Cyclophosphamide (C).

Secondary objectives will investigate duration of response (DOR), progression-free survival (PFS) and overall survival (OS) and the safety of the study regimen.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Patients with locally advanced or metastatic, histologically documented TNBC (absence of human epidermal growth factor 2 [HER2], estrogen receptor [ER], and progesterone receptor [PR] expression) PD-L1+ (Immune Cell >1% using Ventana SP142 assay), not amenable to surgical therapy
* Locally advanced or metastatic TNBC, who have received an anti-PD-1/PD-L1 containing regimen in the neoadjuvant/adjuvant setting
* No prior chemotherapy or targeted systemic therapy (including endocrine therapy) or immunotherapy for inoperable locally advanced or metastatic TNBC
* Tissue accessible for biopsies
* Expected survival of > 3 months
* Female or male subject ≥18 years
* Have measurable/evaluable metastatic disease (RECIST 1.1 criteria)
* Performance status 0-1 on Eastern Cooperative Oncology Group Performance Status (ECOG PS)
* Demonstrate adequate organ (kidney, liver) function

Exclusion Criteria:

* Patients with de novo metastatic TNBC OR those who have received 1 or more chemotherapy or targeted systemic therapy (including endocrine therapy) or immunotherapy regimens for advanced disease
* Immunodeficiency or systemic steroid therapy/immunosuppressive therapy within 7 days prior to study entry
* Known history of active Bacillus Tuberculosis (TBC)
* Hypersensitivity to anti- PD-L1 antibodies or its excipients
* Active autoimmune disease
* Known history of non-infectious pneumonitis
* Active infection requiring systemic therapy
* Known history of Human Immunodeficiency Virus (HIV)
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative])
* Live vaccine within 30 days
* Bone or brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 30 months
  Rate of subjects who achieve either a confirmed Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 30 months
  Interval from treatment initiation to disease progression or death, whichever comes first, or to the last disease assessment for patients alive without progression
Overall survival (OS) | 30 months
  Interval from treatment initiation to death or last known alive date
Duration on response (DoR) | 30 months
  Time between the first documented objective response (CR or PR) and the first documented progression or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Munzone, MD, Principal Investigator — European Istitute of Oncology; Francesco Bertolini, Principal Investigator — European Istitute of Oncology
Locations (4):
- Italy (4):
  - Fondazione IRCCS San Gerardo Dei Tintori, Monza, Monza
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Roma
  - Azienda Sanitaria Locale Br, Brindisi
  - European Institute of Oncology, Milan